CLINICAL TRIAL: NCT02101710
Title: A Randomized, Open-label, One Dose, 2-way Crossover Study to Evaluate the Bioequivalence of Elantan SR* 60 mg in Comparison With Imdur SR* 60 mg Under Fasted and Fed Conditions in Healthy Korean Male Subjects (*Sustained Release)
Brief Title: Pharmacokinetic Properties of Isosorbide-5-mononitrate Under Fasting and Fed Condition in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Korea Co., Ltd. (Industry)
Collaborators: Seoul Pharma Laboratories Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD0001
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Isosorbide 5-mononitrate; Elantan; Imdur; Korean; Healthy
MeSH Terms: interventions — Isosorbide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Elantan SR 60 mg fed (Experimental): Elantan SR 60 mg is orally administered on Day 1 of treatment period 1 for Fed group 2 and on Day 1 of treatment period 2 for Fed group 1.
  Interventions: Drug: Elantan SR 60 mg
- Imdur SR 60 mg fed (Experimental): Imdur SR 60 mg is orally administered on Day 1 of treatment period 1 for Fed group 1 and on Day 1 of treatment period 2 for Fed group 2.
  Interventions: Drug: Imdur SR 60 mg
- Elantan SR 60 mg fasted (Experimental): Elantan SR 60 mg is orally administered on Day 1 of treatment period 1 for Fasted group 2 and on Day 1 of treatment period 2 for Fasted group 1.
  Interventions: Drug: Elantan SR 60 mg
- Imdur SR 60 mg fasted (Experimental): Imdur SR 60 mg is orally administered on Day 1 of treatment period 1 for Fasted group 1 and on Day 1 of treatment period 2 for Fasted group 2.
  Interventions: Drug: Imdur SR 60 mg

INTERVENTIONS:
Drug: Elantan SR 60 mg — * Trade Name: Elantan
  * Active Substance: Isosorbide 5-mononitrate
  * Pharmaceutical form: Tablet
  * Concentration: 60 mg
  * Route of Administration: Oral administration
  Other Names: Isosorbide 5-mononitrate
  Arms: Elantan SR 60 mg fasted; Elantan SR 60 mg fed
Drug: Imdur SR 60 mg — * Trade Name: Elantan
  * Active Substance: Isosorbide 5-mononitrate
  * Pharmaceutical form: Tablet
  * Concentration: 60 mg
  * Route of Administration: Oral administration
  Other Names: Isosorbide 5-mononitrate
  Arms: Imdur SR 60 mg fasted; Imdur SR 60 mg fed

SUMMARY:
This study it to evaluate the bioequivalence of Elantan SR 60 mg compared to Imdur SR 60 mg in sixty healthy Korean male subjects.

DETAILED DESCRIPTION:
This study is to evaluate the bioequivalence of Elantan SR 60 mg compared to Imdur SR 60 mg in sixty healthy Korean male subjects. Thirty subjects will be participating in a fasted state and other thirty subjects will be in a fed state. Elantan SR 60 mg and Imdur 60 mg are two formulations of Isosorbide 5-mononitrate.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent is signed and dated by the subject
* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete the schedule of study assessment), visit schedule or medication intake according to the judgment of the investigator
* Subject is healthy Korean male, 19-55 years of age
* Subject is of normal body weight as determined by a body mass index between 18.5 kg/m^2 and 24.9 kg/m^2
* Sitting blood pressure within the following range: SBP (Systolic Blood Pressure), 90-139 mmHg; DBP (Diastolic Blood Pressure ), 50-89 mmHg
* Subject has no abnormal symptom in a physical examination without congenital or chronic disease

Exclusion Criteria:

* Subject has previously participated in this study or subject has previously been assigned to treatment in a study of the medication under investigation in this study
* Subject has participated in another study of an investigational medication (or a medical device) within the last 90 days or is currently participating in another study of an investigational medication (or a medical device)
* Subject has a history of chronic alcohol or drug abuse within the last 6 months
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has a known hypersensitivity to nitrate or to any components of the investigational medicinal product or reference drugs as stated in this protocol
* Subject has the history or present condition of cardiovascular diseases, like acute circulatory failure (shock, vascular collapse), very low BP, acute myocardial infarction with low filling pressures, arrhythmia, left heart failure with low filling pressures, hypotension, acute attacks of angina, constrictive pericarditis, hypertrophic obstructive cardiomyopathy, cardiac tamponade, aortic valve and/or mitral valve stenosis
* Subject has the history or present condition of severe anemia, head trauma, cerebral haemorrhage, hematopenia, severe cerebrovascular insufficiency, glaucoma, gastrointestinal disorder, neurological abnormalities, hepatic disorder, renal, pulmonary or metabolic diseases
* Subject use a phosphodiesterase 5 inhibitor (sildenafil, tadalafil and vardenafil)
* Symptomatic or asymptomatic orthostatic hypotension at screening defined as a 20 mmHg or more decrease in systolic pressure, or 10 mmHg or more decrease in diastolic pressure after 1 and 3 minutes standing with the arm relaxed at the side (time zero begins after the subject is upright). 5 minutes of supine rest is used as baseline
* Subject has the family or personal history of abnormal bleeding
* Subject had clinically relevant out of range values for hematology and clinical chemistry parameters. However, in agreement with the sponsor, the Investigator may include a subject having values outside the accepted range if, in his/her opinion, these values are of no clinical significance and justification is given
* Subject had any clinically relevant abnormality in physical examination
* Subject has made a blood donation or had a comparable blood loss (>400ml) within the last 3 months prior to the first day of dosing
* Any clinical conditions that in the opinion of the Investigator would make the subject unsuitable for the study
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption due to the presence of lactose
* Subjects who have taken drug products that are enzyme inducers, such as barbiturates, or inhibitors; or who drank excessive alcohol within one month prior to the initiation of the BE (Bioequivalence) study
* Subjects who have taken drug products that could influence the results of the BE study within 10 days before the initiation of the BE study

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve vs. time curve observed from time Baseline to the Last Quantifiable point (AUC(0-t)) | Samples will be taken predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Maximum Observed Plasma Concentration (Cmax) | Samples will be taken predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to infinity (AUC(0-inf)) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Time to reach a maximum plasma concentration (tmax) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Terminal half-life (t1/2) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Rate constant of elimination (λz) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Apparent total body clearance (CL/f) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Apparent volume of distribution (Vz/F) | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
AUC % extrapolation | Samples will be taken 0 (predose) and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 and 36 hr post-dose
Percentage of subjects with at least one Treatment-emergent Adverse Event (TEAE) from the Day 1 of the first treatment period until Safety Follow Up visit | From the Day 1 of the first treatment period until Safety Follow Up visit (Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (1):
- 1, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Jin C, Jeon JY, Im YJ, Jeong JA, Kim Y, Chae SW, Bentz J, Kumke T, Kim MG. Pharmacokinetic properties of isosorbide-5-mononitrate under fasting and fed conditions in healthy male subjects. Int J Clin Pharmacol Ther. 2015 Jan;53(1):97-106. doi: 10.5414/CP202169. PMID 25492848